CLINICAL TRIAL: NCT04823455
Title: Results Following Fresh-frozen Humeral Head Osteochondral Allograft Reconstruction for Reverse Hill-Sachs Lesion
Acronym: ALLO-OMERO2020
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Istituto Ortopedico Rizzoli (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: ALLO-OMERO
Record Dates: First submitted 2021-03-29; First posted 2021-03-30 (Actual); Last update posted 2024-09-23 (Actual); Status verified 2024-09

CONDITIONS: Shoulder Dislocation Closed Traumatic
Keywords: shoulder dislocation, humeral allograft, locked posterior dislocation
MeSH Terms: conditions — Shoulder Dislocation

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Allo Omero 2020 (Experimental): Humeral allograft group 12 patients were surgically treated for a locked posterior glenohumeral dislocation with a humeral head defect affecting at least 30% of the head diameter. During surgery, the bone defect was substituted with a fresh-frozen humeral head osteochondral allograft.Included patients were clinically and radiographically re-evaluated for the purpose of this study by examiners not involved in the primary treatment at a mean of 66 months postoperatively. The clinical examination consisted of a physical examination and structured interview. Computed tomography (CT) was carried out at the medium follow-up of 66 months in all patients to evaluate OA progression and allograft resorption.
  Interventions: Procedure: fresh-frozen humeral head osteochondral allograft reconstruction for reverse Hill-Sachs lesion

INTERVENTIONS:
Procedure: fresh-frozen humeral head osteochondral allograft reconstruction for reverse Hill-Sachs lesion — Between 2001 and 2018, a total of 12 consecutive patients were surgically treated for a locked posterior glenohumeral dislocation with a humeral head defect affecting at least 30% of the head diameter. During surgery, the bone defect was substituted with a fresh-frozen humeral head osteochondral allograft.

SUMMARY:
Locked posterior glenohumeral dislocations with a reverse Hill-Sachs impaction fracture involving less than 30% of the humeral head are most frequently treated with lesser tuberosity transfer into the defect, whereas those involving more than 50% undergo humeral head arthroplasty. Reconstruction of the defect with segmental femoral osteochondral allografts has been proposed to treat patients between these two ranges, but the medium-/long-term outcomes of this joint-preserving procedure are controversial.

DETAILED DESCRIPTION:
Twelve patients with a unilateral locked posterior shoulder dislocation and at least 30% (mean 31%) impaction of the humeral head were treated with segmental reconstruction of the defect with fresh-frozen humeral head osteochondral allografts. Patients were assessed clinically, radiographically and with computed tomography (CT) at a medium follow-up of 66 months (range, 24-225).All twelve shoulders presented a slight limitation in anterior elevation

ELIGIBILITY:
Inclusion Criteria:

- Diagnosis of an acute non-reducible posterior gleno-humeral dislocation with an associated McLaughlin lesion affecting more than 30% of the cartilaginous circumference of the humeral head.

Exclusion Criteria:

- Patients with associated injuries to the affected upper limb, with neuromuscular or psychomotor disorders or with disorders affecting connective tissues.

Ages: 18 Years to 90 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 12 (Actual)
Dates: Start 2020-06-05 (Actual); Primary Completion 2020-08-05 (Actual); Study Completion 2021-04-30 (Actual)

PRIMARY OUTCOMES:
Western Ontario Shoulder Instability index (WOSI) | 2 months
  The WOSI score questionnaire is a tool designed for self-assessment of shoulder function for patients with instability problems.
  Overall scores range from 0 to 2100 with a score of 0 indicating better shoulder function and 2100 indicating worse shoulder function.
American Shoulder and Elbow Surgeons Shoulder Score (ASES) | 2 months
  The American Shoulder and Elbow Surgeons Shoulder Score (ASES) was designed to assess the condition of the shoulder, regardless of disease pathology.
  The ASES is a composite instrument, requiring both a physician assessment and a patient-completed portion; however, it is commonly presented as solely the patient-reported survey. This includes a section on pain (7 items) and a section on activities of daily living (10 items). Scores range from 0 to 100 with a score of 0 indicating a worse shoulder condition and 100 indicating a better shoulder condition.
Constant-Murley score (CS) | 2 months
  The Constant-Murley score is a 100-points scale composed of a number of individual parameters. These parameters define the level of pain and the ability to carry out the normal daily activities of the patient.The Constant-Murley score was introduced to determine the functionality after the treatment of a shoulder injury. The test is divided into four subscales: pain (15 points), activities of daily living (20 points), strength (25 points) and range of motion: forward elevation, external rotation, abduction and internal rotation of the shoulder (40 points). The higher the score, the higher the quality of the function.

SECONDARY OUTCOMES:
Samilson-Prieto score | 2 months
  The Samilson-Prieto classification system is based on the presence and size of osteophytes and the rate of arthrosis in the uninvolved shoulder reflects the high sensitivity of this system. The prevalence of arthritis is often reported in long-term follow-ups after trauma or surgery.
  The higher the score, the worse the arthritis.

CONTACTS AND LOCATIONS:
Locations (1):
- IRCCS Istituto Ortopedico Rizzoli, Bologna, Italy

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Marcheggiani Muccioli GM, Rinaldi VG, Lullini G, Ritali A, Mosca M, Romagnoli M, Guerra E, Zaffagnini S. Mid-Term outcomes following fresh-frozen humeral head osteochondral allograft reconstruction for reverse Hill Sachs lesion: a case series. BMC Musculoskelet Disord. 2021 Sep 8;22(1):768. doi: 10.1186/s12891-021-04657-z. PMID 34496807